CLINICAL TRIAL: NCT00598429
Title: Randomized Clinical Trial of Inhaled PGE1 (IPGE1) in Neonatal Hypoxemic Respiratory Failure. A Protocol for the NICHD Neonatal Research Network
Brief Title: Inhaled PGE1 in Neonatal Hypoxemic Respiratory Failure
Acronym: IPGE1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to lack of recruitment
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0037; U10HD036790 (NIH); U10HD021364 (NIH); U10HD021385 (NIH); U10HD027880 (NIH); U10HD034216 (NIH); U10HD040492 (NIH); U10HD040689 (NIH); U10HD053089 (NIH); U10HD053109 (NIH); U10HD053119 (NIH); U10HD053124 (NIH)
Record Dates: First submitted 2008-01-10; First posted 2008-01-21 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2015-07

CONDITIONS: Infant, Newborn; Respiratory Insufficiency; Pulmonary Hypertension; Respiratory Distress Syndrome, Newborn; Streptococcal Infections
Keywords: NICHD Neonatal Research Network; Hypoxemic respiratory failure (HRF); Persistent pulmonary hypertension of the newborn (PPHN); Prostaglandin E1 (PGE1); Mechanical ventilation; Meconium, aspiration
MeSH Terms: conditions — Respiratory Insufficiency; Hypertension, Pulmonary; Respiratory Distress Syndrome, Newborn; Streptococcal Infections; Persistent Fetal Circulation Syndrome; Meconium Aspiration Syndrome | interventions — Alprostadil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High dose (Active Comparator): PGE1 300 ng/kg/min via nebulizer over a 72-hour period
  Interventions: Drug: Inhaled Prostaglandin E1
- Low dose (Active Comparator): PGE1 150 ng/kg/min via nebulizer over a 72-hour period
  Interventions: Drug: Inhaled Prostaglandin E1
- Placebo (Placebo Comparator): Normal saline, the diluent for the drug, via nebulizer over a 72-hour period
  Interventions: Drug: Inhaled Prostaglandin E1

INTERVENTIONS:
Drug: Inhaled Prostaglandin E1 — Delivery of one dose of either high dose PGE1 (300 ng/kg/min), low dose PGE1 (150 ng/kg/min), or placebo (normal saline, the diluent for the drug) via nebulizer over a 72-hour period
  Other Names: Alprostadil

SUMMARY:
This pilot study was a randomized, placebo-controlled, clinical trial to test the safety of using the intravenous form of Prostaglandin E1 (PGE1) in an inhaled form for treatment of hypoxemic respiratory failure in term newborns. The study planned to enroll 50 infants diagnosed with hypoxemic respiratory failure at nine NICHD Neonatal Research Network sites, and randomly assign them to receive one dose over a 72-hour period of either high concentration PGE1 (300 ng/kg/min), low concentration PGE1 (150 ng/kg/min), or placebo (normal saline, the diluent for the drug). In addition to determining the safety, optimal dose, and duration of the therapy, this pilot trial planned to evaluate the feasibility of conducting a larger, multi-center randomized, blinded placebo-controlled trial.

DETAILED DESCRIPTION:
Hypoxemic respiratory failure (HRF), frequently associated with persistent pulmonary hypertension of the newborn (PPHN), is a rare, but life-threatening condition affecting approximately 2 to 9 percent of infants admitted to neonatal intensive care units and results in significant morbidity and mortality. It occurs more often in full- or post-term babies whose circulatory systems do not adapt well to breathing outside the womb. HRF may result from congenital hernia of the diaphragm, group B streptococcal infection, inhaling meconium in the womb, or respiratory distress syndrome.

Medical treatments, such as high frequency ventilation, inhaled nitric oxide, and Extracorporeal Membrane Oxygenation (ECMO, a heart and lung support machine), have significantly increased survival of children with HRF. These therapies, while successful, however, have a variety of side effects and potential long-term disabilities.

This feasibility trial was designed to test the safety of using the intravenous form of Prostaglandin E1 in an inhaled form (iPGE1) on infants born at 34 0/7ths weeks gestational age or greater diagnosed with hypoxemic respiratory failure and on assisted ventilation. The intravenous form of PGE1 was to be aerosolized and administered via a nebulizer attached to the infant's ventilator. The goal was to enroll 50 subjects within 6-9 months, in preparation for a larger, multi-center randomized control trial; however, the study was withdrawn for lack of recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at 34 0/7ths weeks gestational age or greater (by best obstetrical estimate) and at a postnatal age no greater than 7 days (168 hours)
* Infants diagnosed with hypoxemic respiratory failure (HRF), including perinatal aspiration syndrome (meconium, blood, or amniotic fluid), pneumonia/ sepsis, respiratory distress syndrome, or idiopathic respiratory failure
* Infants who will receive assisted ventilation for HRF
* Infants with an oxygenation index (MAP x FiO2 x 100/PaO2)(OI) of 15-25 on two arterial gases taken between 15 minutes and 12 hours apart
* An indwelling arterial line
* Infants whose parents/legal guardians have provided consent for enrollment

Exclusion Criteria:

* Any infant in whom a decision has been made not to provide full treatment
* Known structural congenital heart disease, except patent ductus arteriosus and atrial/ventricular level shunts
* Congenital diaphragmatic hernia
* Preterm neonates less than 34 weeks
* Thrombocytopenia (platelet count < 80,000/μl) unresponsive to platelet transfusion
* Infants receiving hypothermia for hypoxic ischemic encephalopathy
* Previous treatment with inhaled nitric oxide
* Infants already enrolled in a conflicting and/or Investigational New Drug (IND) clinical trial
* Infants whose parents/legal guardians refuse consent

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The ability to recruit an adequate number of patients (n = 50) in a 6-9 month period without excessive (>20%) protocol violations. | 6-9 months after trial begins recruitment

SECONDARY OUTCOMES:
Progression to an OI greater than 25 | 72-hours after enrollment
Improvement in partial pressure of oxygen (PaO2) in the blood gas | 72-hours after enrollment
Change in OI | 72 hours after enrollment
Death | 72-hours after intervention
Need for inhaled nitric oxide or ECMO | 72-hours after enrollment
Length of hospitalization
Duration of mechanical ventilation
Number of days of oxygen used and need for supplemental oxygen at 28 days of life
Occurrence of grade III-IV intracranial hemorrhage and cystic leukomalacia

CONTACTS AND LOCATIONS:
Overall Officials: Michele C. Walsh, MD MS, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Ronald N. Goldberg, MD, Principal Investigator — Duke University; Krisa P. Van Meurs, MD, Principal Investigator — Stanford University; Ivan D. Frantz III, MD, Principal Investigator — Tufts Medical Center; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Edward F. Bell, MD, Principal Investigator — University of Iowa; Kristi L. Watterberg, MD, Principal Investigator — University of New Mexico; Roger G. Faix, MD, Principal Investigator — University of Utah; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Pablo J. Sanchez, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - University of Iowa, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Sood BG, Keszler M, Garg M, Klein JM, Ohls R, Ambalavanan N, Cotten CM, Malian M, Sanchez PJ, Lakshminrusimha S, Nelin LD, Van Meurs KP, Bara R, Saha S, Das A, Wallace D, Higgins RD, Shankaran S; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Inhaled PGE1 in neonates with hypoxemic respiratory failure: two pilot feasibility randomized clinical trials. Trials. 2014 Dec 12;15:486. doi: 10.1186/1745-6215-15-486. PMID 25496504
- See also: NICHD Neonatal Research Network — https://neonatal.rti.org/